CLINICAL TRIAL: NCT06814522
Title: Psilocybin-Assisted Therapy for Physician Well-Being and Burnout: Feasibility, Safety, Clinical Effectiveness and Biomarkers of Response [PAT-B (Psilocybin-Assisted Therapy for Physician Well-Being and Burnout)]
Brief Title: Psilocybin-Assisted Therapy for Physician Well-Being and Burnout
Acronym: PAT-B
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Cory Weissman, Dr. Cory Weissman, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 176596
Record Dates: First submitted 2025-02-01; First posted 2025-02-07 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Burnout; Burnout, Healthcare Workers
Keywords: burnout; physician; doctor
MeSH Terms: conditions — Burnout, Psychological | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psilocybin-Assisted Therapy (Experimental): Subjects will receive a single dose of psilocybin in conjunction with psychedelic-assisted therapy.
  Interventions: Drug: Psilocybin, [3-[2-(dimethylamino)ethyl]-1H-indol-4-yl] dihydrogen phosphate

INTERVENTIONS:
Drug: Psilocybin, [3-[2-(dimethylamino)ethyl]-1H-indol-4-yl] dihydrogen phosphate — 25 mg, single dose of psilocybin
  Other Names: Psilocybin

SUMMARY:
Through an open-label study involving a small group of UCSD physicians experiencing burnout, the investigators will evaluate the feasibility, safety, and preliminary effectiveness of PAT to reduce burnout symptoms.

DETAILED DESCRIPTION:
Physician burnout is a critical issue. Research shows that physician burnout is increasing, that physicians suffer higher rates of burnout than the general population, and that physician burnout is associated with poor mental health outcomes.

Psilocybin is a naturally occurring alkaloid within certain fungi that elicits acute perceptual, cognitive, and emotional changes when ingested, due to action on neurotransmitter and neurocirculatory systems. The combination of psilocybin with psychological support, termed Psilocybin-Assisted Therapy (PAT), is a promising new mental health intervention shown to produce rapid and sustained improvements in psychological domains affected in burnout. PAT demonstrates preliminary efficacy as a treatment for depression and substance use disorders, is associated with brain changes measured with electroencephalography (EEG) and is a strong candidate treatment for physician burnout.

The primary aim of this study is to investigate the safety, feasibility, and preliminary efficacy of PAT to enhance well-being in University of California, San Diego (UCSD) physicians experiencing burnout. A secondary aim is to identify neurophysiological changes associated with response to PAT. Physicians experiencing burnout will be recruited in an open-label trial involving preparatory therapy sessions, psilocybin treatment, and post-treatment integration. Burnout will be measured with the Stanford Professional Fulfillment Index (PFI).

ELIGIBILITY:
Inclusion Criteria:

1. UCSD faculty physician, aged 21-70. Volunteer faculty are not included
2. Meets criteria for physician burnout
3. Experiencing symptoms of burnout for >6 months
4. Able to complete all required study visits
5. Not previously diagnosed with a serious mental illness (including schizophrenia, bipolar disorder, and severe depression), or substance use disorder as confirmed in clinical interview
6. Not currently taking any psychotropic medications or nonpsychotropic medication that may be associated with serotonin syndrome, such as serotonin reuptake inhibitors (SSRI or SNRI), dextromethorphan, linezolid, tramadol, meperidine

Exclusion Criteria:

1. Previous inpatient psychiatric hospitalization(s)
2. Previously diagnosed with a psychotic disorder (schizophrenia, schizoaffective disorder, or other psychotic spectrum disorder), bipolar spectrum disorder, personality disorder (borderline personality disorder, antisocial personality disorder, or other severe personality disorders), any severe psychiatric disorder.
3. Exhibiting elevated suicide risk
4. First degree family history of psychosis or bipolar disorder
5. Prior exposure to psilocybin or other psychedelic compounds in the previous 10 years
6. Currently pregnant, nursing, planning pregnancy, engaging in sexual intercourse without effective contraceptive method in last three months
7. Those who plan to donate sperm within three months following the study.
8. Known cardiovascular disease including history of stroke, myocardial infarction, uncontrolled hypertension, valvular heart disease, tachycardia, elongated QT interval, or clinically significant arrythmia.
9. History of seizure disorder
10. Use of recreational illicit drugs
11. Clinically concerning results from vital signs, ECG, physical examination, or laboratory tests during screening
12. Any other clinically significant illnesses deemed to pose risk for the participant

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Stanford Professional Fulfillment Index (PFI) | From enrollment until end of study at 12 week follow-up.
  Assessment used to determine degree/severity of burnout.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No